CLINICAL TRIAL: NCT02848573
Title: the Correlation Between Hepatic Fibrotic Scores and ADC and Other Non-invasive Indicators in Patients With Biliary Atresia
Brief Title: the Correlation Between Non-invasive Indicators in Patients With Biliary Atresia
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Assistant Professor, National Taiwan University Hospital
Other Study IDs: 201403098RINC
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: to Find Out Non-invasive Indices to Predict the Status of Hepatic Fibrosis in BA Patients.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
we propose this study and try to find out possible clinical applicable non-invasive imaging indices or its combination with the laboratory indices to predict the status of hepatic fibrosis in BA patients.

ELIGIBILITY:
Inclusion Criteria:

* pathological proved diagnosis of biliary atresia, and without other distinct abnormality or malformations. All had undergone Kasai portoenterostomy. All of them received abdominal MRI study.

Exclusion Criteria:

* absence of laboratory data required.

Ages: 10 Days to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: biliary atresia
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-04; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
pathologic METAVIR fibrosis score | 1 month